CLINICAL TRIAL: NCT02497209
Title: International AGD Database; Determinants of AGD and Establishment of Normative Data
Acronym: iAGD
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Anders Juul, Professor, Rigshospitalet, Denmark
Other Study IDs: AGD5064
Record Dates: First submitted 2015-07-10; First posted 2015-07-14 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Decreased Anogenital Distance

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: No

SUMMARY:
Aim: To collate data on Anogenital Distance (AGD) from several population studies to build an international database for Anogenital Distance (AGD) Primary objective: To build a database platform to promote and facilitate international collaboration on research related to AGD, endocrine disruptors and reproductive health.

Study Design Observational study Outcome Measures Outcomes from varying projects based on the database

Summary of eligibility criteria Population studies with subjects in whom data on AGD is available

Procedures:

An international AGD database will be set-up with an appropriate dataset for the research projects. This will be based on anonymised data from multiple population studies. In order to facilitate and provide a governance structure for the study, an international AGD consortium will be established.

DETAILED DESCRIPTION:
Introduction Increasing incidence of cryptorchidism, hypospadias, and testicular cancer has paralleled the concomitant decline in male fertility in several countries(1). Exposures of environmental agents, which act as endocrine disruptors resulting in abnormalities in the development and function of fetal tests, have been hypothesised to underlie these trends. However, these outcomes are relatively rare, and in some cases occur a long period after exposure. Development of a sensitive biomarker of fetal androgen action during infancy is critical to evaluate the effects of potential endocrine disrupting environmental agents on the reproductive system.

Anogenital distance (AGD) defined as the distance from the anus to genital tubercle is a sensitive marker for prenatal exposure to endocrine-disrupting chemicals in animals (1,2). However, unlike in animals, the external genitalia are well differentiated in humans and the anatomical landmarks to measure AGD have been a matter of debate. This has resulted in several proxy measurements of AGD using multiple anterior landmarks such as anterior insertion of the penis, posterior insertion of penis or perineoscrotal junction (3).

Nevertheless, several human studies have reported an association between exposure to a variety of commonly used environmental chemicals and reduction in AGD in humans (1,2,4). AGD remains the single biomarker, which has showed consistent alterations related to prenatal exposure to environmental agents with established endocrine-disrupting activity in animals. Furthermore, a reduced AGD has been shown in common disorders of male reproductive health such as hypospadias, cryptorchidism, reduced semen quality and infertility (1,2,5).

Rationale for the study The use of AGD in epidemiological studies has several limitations. Varying methods used for measurement is believed to result in considerable variations in the AGD values (6). A few small studies have also suggested the possibility of ethnic variation. Normative data is vital particularly in cross-sectional studies. Normative data for some types of AGD has been published, however, population data using more standardised methods for measurement and on other types of AGD are vital in understanding the potential effect of endocrine disruptors on reproductive health (7,8). Large datasets from international collaboration are important to study variations related to types of measurement techniques and ethnicity, and explore the relationship between AGD, environmental exposures and male reproductive disorders.

The aim of the project is to set up an international AGD database to promote and facilitate research in the area related to AGD and, therefore, provide the researchers access to a large dataset derived from multiple studies.

Study Design Cohorts of healthy subjects from populationbased studies which included measurements of anogenital distance will be included.

International AGD database An international AGD database (IAGD) will be established and located in the Department of Growth and Reproduction, Rigshospitalet, Copenhagen, Denmark. The database will consist of anonymised data from multiple studies. For each approved research project, appropriate data will be exported from the contributing studies to the international database.

International AGD Consortium An international AGD consortium will provide the governance framework for the international AGD database. This consortium will consist of the founding members and a member from each of the contributing studies. They will be responsible for advising on the design and structure of the database, evaluating and approving specific research projects.

Database management & Data Protection For each research project approved by the consortium, the members (PI's of the contributing studies) will be asked for permission for their data to be included. The data relevant for each specific research project will be extracted from the contributing studies, which expressed an interest in the project and exported to the international AGD database. This database will be unlinked from the original databases for the participating studies so that subjects will not be identified by linkage. The data will be anonymised, and no patient identifiable information including the date of birth will be exported to the international database. Furthermore, no data, which could potentially link international AGD database with that of the contributing studies such as the study specific identifier for the contributing study, will be exported to the international database.

In addition, the database will have relevant details of all the contributing studies including participant numbers, the schedule of assessments and collection of biological samples, and method of measurements.

Ethical & Regulatory considerations

International AGD database The database will be located in Rigshospitalet, Copenhagen, Denmark and comply with Data protection guidance in Denmark. Appropriate regulatory approvals will be obtained from the Data protection agency in Denmark.

Regulatory approvals for the contributing studies The regulatory framework for sharing data with external researchers varies considerably in different countries. Regulatory permissions if necessary will be obtained by the PI's of the contributing studies to share anonymised data with the international database.

Sponsorship & Funding The database will be sponsored by Rigshospitalet, Copenhagen, Denmark. The study will be funded by International Center for Research and Research Training in Endocrine Disrupting Effects on Male Reproduction and Child Health (EDMaRC).

An international Anogenital Distance (AGD) consortium was set up to manage the database. The current members of the consortium are:

Chief Investigators

1. Professor Anders Juul Leader of EDMaRC, Professor, head of department EDMaRC and Department of Growth and Reproduction Rigshospitalet, Copenhagen, Denmark
2. Professor Shanna H Swan Professor and Vice Chair for Research and Mentoring, Department of Preventive Medicine, Mount Sinai Medical Center, NY, NY, USA

   Study management group
3. Dr. Ajay Thankamony Clinical Fellow and Honorary Consultant Department of Paediatrics Cambridge University Hospital, Cambridge UK
4. Professor Katharina M Main Department of Growth and Reproduction Rigshospitalet, Copenhagen, Denmark
5. Dr. Marie Lindhardt Johansen Department of Growth and Reproduction Rigshospitalet, Copenhagen, Denmark
6. Jørgen Holm Petersen Statistician, Department of Growth and Reproduction Rigshospitalet, Copenhagen, Denmark
7. Jørgen Riis Christensen Database Manager, Department of Growth and Reproduction Rigshospitalet, Copenhagen, Denmark
8. Principal investigators of contributing studies

References

1. Juul A, Almstrup K, Andersson A-M, Jensen TK, Jorgensen N, Main KM, Meyts ER-D, Toppari J, Skakkebaek NE 2014 Possible fetal determinants of male infertility. Nat Rev Endocrinol 10:553-562
2. Dean A, Sharpe RM 2013 Anogenital distance or digit length ratio as measures of fetal androgen exposure: relationship to male reproductive development and its disorders. J Clin Endocrinol Metab 98:2230-2238
3. Hsieh MH, Breyer BN, Eisenberg ML, Baskin LS 2008 Associations among hypospadias, cryptorchidism, anogenital distance, and endocrine disruption. CurrUrolRep 9:137-142
4. Swan SH 2006 Prenatal phthalate exposure and anogenital distance in male infants. Environ Health Perspect 114:A88-89
5. Mendiola J, Stahlhut RW, Jorgensen N, Liu F, Swan SH 2011 Shorter anogenital distance predicts poorer semen quality in young men in Rochester, New York. Environ Health Perspect 119:958-963
6. Sathyanarayana S, Grady R, Redmon JB, Ivicek K, Barrett E, Janssen S, Nguyen R, Swan SH 2015 Anogenital distance and penile width measurements in The Infant Development and the Environment Study (TIDES): Methods and predictors. J Pediatr Urol 11:76.e71-76
7. Thankamony A, Ong KK, Dunger DB, Acerini CL, Hughes IA 2009 Anogenital Distance from Birth to Two Years: a Population Study. EnvironHealth Perspect 117:1786-1790
8. Sathyanarayana S, Grady R, Redmon JB, Ivicek K, Barrett E, Janssen S, Nguyen R, Swan SH 2015 Anogenital distance and penile width measurements in The Infant Development and the Environment Study (TIDES): Methods and predictors. J Pediatr Urol

ELIGIBILITY:
Inclusion Criteria:

* subjects from populationbased cohort studies measuring AGD

Exclusion Criteria:

* none

Max Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: An international AGD database (IAGD) will be established and located in the Department of Growth and Reproduction and EDMaRC, Rigshospitalet, Copenhagen, Denmark. The database will consist of anonymised data from multiple studies. For each approved research project, appropriate data will be exported from the contributing studies to the international database.
  International AGD Consortium An international AGD consortium will provide the governance framework for the international AGD database. This consortium will consist of the founding members and a member from each of the contributing studies. They will be responsible for advising on the design and structure of the database, evaluating and approving specific research projects.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2015-08; Primary Completion 2016-12 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Measurement of Anogenital Distance ( AGD) (in milimeter) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Anders Juul, prof, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- EDMaRC, Rigshospitalet secton 5064, Copenhagen, Denmark

REFERENCES:
- [Derived] Fischer MB, Ljubicic ML, Hagen CP, Thankamony A, Ong K, Hughes I, Jensen TK, Main KM, Petersen JH, Busch AS, Upners EN, Sathyanarayana S, Swan SH, Juul A. Anogenital Distance in Healthy Infants: Method-, Age- and Sex-related Reference Ranges. J Clin Endocrinol Metab. 2020 Sep 1;105(9):2996-3004. doi: 10.1210/clinem/dgaa393. PMID 32574349